CLINICAL TRIAL: NCT06663332
Title: A Phase 3, Multicenter, Open-label, Basket, LTE Study to Evaluate the Safety of Guselkumab in Pediatric Participants With Crohn's Disease, Ulcerative Colitis, or Juvenile Psoriatic Arthritis
Brief Title: A Long-term Extension (LTE) Study of Guselkumab in Pediatric Participants
Acronym: TRILOGY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CNTO1959ISD3001; CNTO1959ISD3001 (Other: Janssen Research & Development, LLC); 2023-509560-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohns Disease; Colitis, Ulcerative; Arthritis, Psoriatic; Arthritis, Juvenile
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Psoriatic; Arthritis, Juvenile | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guselkumab (Every 8 weeks) (Experimental): Participants treated with guselkumab in one of the three primary studies (CNTO1959PUC3001 [NCT06260163], CNTO1959PBCRD3007 [NCT05923073], CNTO1275JPA3001 [NCT05083182]) will be enrolled in this long-term extension (LTE) study, if in investigator's opinion, participant will benefit from continued guselkumab therapy and will have continued access to guselkumab (every 8 weeks [q8w]). Participants coming from double-blinded arm of primary studies CNTO1959PUC3001 and CNTO1959PBCRD3007 will be assigned to q8w dosing. Based on investigator's discretion and participant's clinical status, they have option to switch to q4w once during LTE study prior to unblinding of primary study assignment. Once the primary study is unblinded, dosing frequency may be adjusted to match what the participant had received before enrolling in LTE study. Participants coming from study CNTO1275JPA3001 will continue same dosing regimen from primary study (q8w) and cannot change their dosing interval during LTE study.
  Interventions: Drug: Guselkumab
- Guselkumab (Every 4 weeks) (Experimental): Participants treated with guselkumab in one of the three primary studies (CNTO1959PUC3001 [NCT06260163], CNTO1959PBCRD3007 [NCT05923073], CNTO1275JPA3001 [NCT05083182]) will be enrolled in this LTE study, if in the investigator's opinion, the participant will benefit from continued guselkumab therapy. Participants will have continued access to guselkumab (q4w). Participants coming from the open-label arm of the primary studies CNTO1959PUC3001 and CNTO1959PBCRD3007 will be assigned to q4w dosing. No dose adjustments are permitted. Participants coming from the jPsA primary study (CNTO1275JPA3001) will continue the same dosing regimen from the primary study (q4w) and cannot change their dosing interval during the LTE study.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Other Names: CNTO1959

SUMMARY:
The purpose of this study is to evaluate long-term safety of subcutaneous guselkumab in pediatric participants with moderately to severely active ulcerative colitis, or moderately to severely active Crohn's disease, or juvenile psoriatic arthritis (jPsA).

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the dosing planned in the primary pediatric guselkumab study
* Must have received benefit from continued guselkumab therapy in the opinion of the investigator
* Before enrollment, a participant must be either: (a) Not of childbearing potential, OR (b) Of childbearing potential and not sexually active, practicing abstinence or a highly effective method of contraception and agrees to remain on a highly effective method while receiving study intervention and until 12 weeks after the last dose - the end of relevant systemic exposure
* Parent(s) (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study. Assent is required from participants who are capable of understanding the nature of the study, typically those aged 7 years and older, to ensure their willingness to participate. An adolescent who provides assent will have the opportunity to sign an adult ICF upon reaching the age of majority, thereby affirming their understanding of the study's purpose and procedures, as well as their willingness to participate.

Exclusion Criteria:

* Participant is greater than or equal to (>=) 18 years of age and resides in a country where 2 years have elapsed post marketing authorization for the respective adult indication
* Participant is <18 years of age and resides in a county where 2 years have elapsed post marketing authorization for the respective pediatric indication
* Are pregnant, nursing, or planning pregnancy or fathering a child
* Have taken any disallowed therapies before the planned first long-term extension (LTE) dose of study intervention
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2031-12-12 (Estimated); Study Completion 2031-12-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events as Assessment of Safety | Up to 6 years and 9 months
  Treatment-emergent adverse events will be reported to analyze the long-term safety of guselkumab in pediatric participants.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
- Instituto Caici, Rosario, Argentina
- China (6):
  - Capital Center For Children's health Capital Medical University, Beijing
  - Changzhou No 2 Peoples Hospital, Changzhou
  - The Childrens Hospital Zhejiang University School Of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
- Schon Klinik Hamburg Eilbek, Hamburg, Germany
- Italy (2):
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - Azienda USL di Bologna - Ospedale Maggiore, Bologna
- Japan (5):
  - Kanazawa University Hospital, Kanazawa
  - Kobe University Hospital, Kobe
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Shinshu University Hospital, Matsumoto
  - Saga University Hospital, Saga
- Poland (3):
  - Centrum Zdrowia Dziecka i Rodziny im Jana Pawla II w Sosnowcu Sp z o o, Sosnowiec
  - Medical Network, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Uls Braga - Hosp. Braga, Braga, Portugal
- Samsung Medical Center, Seoul, South Korea
- Hosp. Clinico Univ. de Santiago, Santiago de Compostela, Spain
- Turkey (Türkiye) (2):
  - Gazi University Medical Faculty, Ankara
  - Umraniye Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency